CLINICAL TRIAL: NCT05302765
Title: Intravenous Fluid Administration's Effect on Pediatric Lumbar Puncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Austin Wheeler, Fellow, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UAB IRB#: IRB-300008761
Record Dates: First submitted 2022-03-17; First posted 2022-03-31 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Lumbar Puncture

STUDY DESIGN:
Intervention Model Description: The control arm consists of lumbar puncture performed in routine fashion without the administration of intravenous fluids prior to procedure. The experimental arm will undergo normal saline intravenous fluids administration (20 milliliters/kilogram) prior to lumbar puncture. Bolus to be complete prior to lumbar puncture in the experimental group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No IV Fluids (No Intervention): The control arm consists of lumbar puncture performed in routine fashion without the administration of intravenous fluids prior to procedure.
- Receives IV Fluids (Experimental): The experimental arm will receive normal saline intravenous fluid administration (20 milliliters/kilogram) prior to lumbar puncture. Bolus to be complete prior to lumbar puncture in the experimental group.
  Interventions: Other: Normal Saline Intravenous Fluids

INTERVENTIONS:
Other: Normal Saline Intravenous Fluids — Administration of normal saline intravenous fluids (20 milliliters/kilogram).
  Arms: Receives IV Fluids

SUMMARY:
The purpose of this project is to determine if administration of normal saline intravenous fluids prior to a lumbar puncture improves first time success of lumbar puncture in infants less than 3 months of age. First time success of lumbar puncture defined as cerebrospinal fluid obtained on the first attempt with less than 1000 red blood cells per mm3 in the fluid specimen.

DETAILED DESCRIPTION:
Lumbar Puncture is a common procedure performed in the Pediatric Emergency Department. This procedure is often performed to assess the cerebrospinal fluid for infection. At Children's of Alabama, approximately 75% of patients undergoing this procedure are ages 3 months of age or younger. There is hypothesis that intravenous fluid administration prior to performing a lumbar puncture in this age group will increase the chances of obtaining non-bloody spinal fluid in less attempts.

A recent study by Rankin et al, infants 0 to 3 months with the diagnosis of pyloric stenosis in a pediatric emergency department were enrolled. This study measured the subarachnoid space in millimeters squared before and 1 hour after administration of normal saline intravenous fluid bolus with the use of ultrasound. The sample size was 40 patients with a mean age of 11.3 days. The study determined that fluid boluses were not associated with a significant increase in the sonographic measurement of the subarachnoid space. However, no lumbar punctures were actually performed in their study. Based on their results, they deduced that fluids may not increase lumbar puncture success rates. No studies have been published evaluating whether intravenous fluids affect the success rate of performed lumbar punctures.

A prospective randomized control trial will be performed with patients of the ages 0 to 3 months. Patients to be enrolled will be all patients 3 months or less in the Children's of Alabama Pediatric Emergency Department who will be undergoing a lumbar puncture procedure as part of their clinical work-up. The control arm will have the lumbar puncture performed in routine fashion without the administration of intravenous fluids prior to procedure. The experimental arm will undergo normal saline intravenous fluids (20 milliliters/kilogram) prior to lumbar puncture. The bolus is to be completed prior to performing the lumbar puncture in the experimental group.

Physicians and Nurse Practitioners caring for patients who are performing a lumbar puncture as part of their clinical work-up are responsible for identifying the patient as a candidate for the study. The providers identifies if patients in the age group are a candidate for enrollment based on inclusion and exclusion criteria.

If the patient is identified to be an acceptable candidate for the study, the provider caring for the patient notifies a physician in the Emergency Department who is qualified to obtain consent for the study. Consents are available in both English and Spanish. Once consent is obtained, providers obtain a sealed packet that contains a randomized assignment into one of the arms of the study. If the patient is assigned to the experimental arm, the provider orders a 20 mL/Kg normal saline intravenous fluid bolus and performs the lumbar puncture after the bolus has completed. If the patient is assigned to the control arm, the provider proceeds with the lumbar puncture without ordering or administering intravenous fluids.

After the lumbar puncture is completed, the provider performing the lumbar puncture fills out a brief data collection form that is kept within the randomization packet. This data form collects information that is not routinely documented within the electronic medical record including medical record number, arm of study (experimental vs control), training level of provider that performed each attempt, specialty of provider that performed each attempt, position of patient during each attempt, and on which attempt, if any, CSF was obtained. These data forms are routinely collected. Chart review is performed using medical record numbers from the data collection form to collect additional information into a de-identified excel data sheet. Data obtained from chart review includes age of patient, gestational age, weight, gender, ethnicity, preferred language, duration from intravenous fluid bolus to collection of cerebrospinal fluid, cerebrospinal fluid appearance, training level of provider who performed the first attempt and final attempt, total number of attempts, position of patient during lumbar puncture, number of red blood cells in cerebrospinal fluid, number of white blood cells in cerebrospinal fluid, protein count in cerebrospinal fluid, glucose in cerebrospinal fluid, additional testing, and reasoning for lumbar puncture.

ELIGIBILITY:
Inclusion Criteria:

* Ages 0 and 3 months
* Patient at Children's of Alabama's Emergency Department
* Undergoing a lumbar puncture as part of their clinical work-up

Exclusion Criteria:

* Vertebral abnormalities
* Severe scoliosis
* Lumbar puncture to be performed by interventional radiology
* Received intravenous fluids prior to study enrollment
* Hypotension requiring fluid resuscitation
* Shock requiring fluid resuscitation
* Ultrasound assistance
* Lumbar puncture performed or attempted at another hospital within 24 hours

Ages: 0 Months to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 182 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Successful Lumbar Puncture | 1 to 1.5 hours
  Cerebrospinal fluid obtained on first attempt with less than 1000 red blood cells per mm3 in fluid.

SECONDARY OUTCOMES:
Successfully Obtaining Cerebrospinal Fluid | 1 to 1.5 hours
  Total number of attempts to obtain cerebrospinal fluid
Time from intravenous fluid bolus completion to cerebrospinal fluid collection | 0 minutes to 1.5 hours
  Time in minutes from bolus completion to CSF collection and it's effect on success rates
Level of trainings effect on successful lumbar punctures | 1 to 1.5 hours
  Outcomes sub-grouped by provider's level of training

CONTACTS AND LOCATIONS:
Locations (1):
- Children's of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rankin J, Wang VJ, Goodarzian F, Lai HA. Intravenous Fluid Bolus Prior to Neonatal and Infant Lumbar Puncture: A Sonographic Assessment of the Subarachnoid Space After Intravenous Fluid Administration. JAMA Pediatr. 2016 Mar;170(3):e154636. doi: 10.1001/jamapediatrics.2015.4636. Epub 2016 Mar 7. PMID 26954534